CLINICAL TRIAL: NCT04615559
Title: Contrast Enhanced Ultrasound Endoleak Identification and Classification Compared to Computed Tomography in High-risk Complicated Aneurysm Repair Patients
Brief Title: Contrast Enhanced Ultrasound Endoleak Identification and Classification
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study team did not proceed with study start-up.
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Edward Grant, Professor of Clinical Radiology, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS-20-00428
Record Dates: First submitted 2020-10-28; First posted 2020-11-04 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- contrast enhanced ultrasound (Experimental): CEUS will be performed at one month post-op, six months post-op and at one year.
  Interventions: Diagnostic Test: Contrast enhanced ultrasound

INTERVENTIONS:
Diagnostic Test: Contrast enhanced ultrasound — CEUS involves the use of microbubble contrast agents and specialized imaging techniques to enhance the signal from blood, thus showing flow in macroscopic vessels as well as tissue perfusion information

SUMMARY:
Surgery for abdominal aortic pathology usually occurs in the setting of advanced cardiovascular disease. The repair can be relatively simple or complex with multiple steps including open repair, placing a stent with a catheter, and placing a complicated stent that allows for crossing vessels without occluding them. All these repairs require imaging follow up. The most commonly accepted tool for follow up is Computed Tomography (CT) scan which involves ionizing radiation and potentially nephrotoxic iodinated contrast. Recommendations for the time interval for follow up, as well the radiology imaging technique vary. Routine ultrasound with Doppler, CT, and MRI has all been employed utilizing various imaging protocols. Clinicians use non-contrast CT, arterial phase and delayed phase CT, ultrasound, and various combinations based on personal experience and patient pathology. Concerns over cost, potential nephrotoxicity of contrast agents and repeated radiation exposure has led to investigation of alternate imaging modalities such as contrast-enhanced ultrasound (CEUS). CEUS represents an improvement of ultrasound imaging but comparisons against CT report widely varying results, likely due to technical factors of CEUS and limitations of single-phase CTA. Contrast ultrasound has been used effectively to diagnose leaks in the aorta post repair and is without the radiation and potential nephrotoxicity of iodinated contrast. Of yet, no large prospective studies have compared CT and contrast US and no studies have looked at the more complicated staged or fenestrated repairs. This study proposes to perform a contrast ultrasound at the same time as a contrast CT using a standardized protocol. This protocol would include a non-contrast CT, angiographic CT, and a CT in a delayed phase in all patients as standard of care. We will compare the results of a contrast US with the various data derived from a three phase CT.

DETAILED DESCRIPTION:
Introduction: Surgery for abdominal aortic pathology usually occurs in the setting of advanced cardiovascular disease. The repair can be relatively simple or complex with multiple steps including open repair, placing a stent with a catheter, and placing a complicated stent that allows for crossing vessels without occluding them. All these repairs require imaging follow up.

Rationale: The most commonly accepted tool for follow up is Computed Tomography (CT) scan which involves ionizing radiation and potentially nephrotoxic iodinated contrast. Routine ultrasound with Doppler, CT, and MRI has all been employed utilizing various imaging protocols. Concerns over cost, potential nephrotoxicity of contrast agents and repeated radiation exposure has led to investigation of alternate imaging modalities such as contrast enhanced ultrasound (CEUS). CEUS also allows continuous (dynamic) or real-time monitoring of the aneurysm and endoleak throughout the study.

Objectives:

Aim 1: To determine the consistency/discrepancy of endoleak detection (positive/negative) for contrast enhanced ultrasound (CEUS) versus various phases of CTA versus delayed phase CTA.

Aim 2 (Exploratory): To explore the consistency/discrepancy of endoleak type (type 1-5) between CEUS and delayed phase CTA.

Aim 3 (Exploratory): To explore the consistency/discrepancy of endoleak source detected (positive/negative for each source) for type II endoleaks between CEUS and CTA.

Aim 4 (Exploratory): Re-assess Aims 1-3 for the follow-up scans. The goal for this aim is to examine whether the consistency/discrepancy patterns discovered in Aims 1-3 can be repeated at the follow-up scans.

Population: 40 patients who have undergone an EVAR or FEVAR for abdominal aortic aneurysms and are expected to have CTA as part of their standard of care will be enrolled in the study.

Methodology: Patients will be evaluated with research contrast ultrasound at one month post-op, six months post-op and at one year.

Data Analysis Plan: Binomial 95% confidence interval will be calculated for sensitivity and specificity. One- sided binomial test will be conducted to test whether the target sensitivity and specificity are superior to the null value, e.g. a minimal acceptable level of sensitivity and specificity. In detecting the rate of endoleak positive on CEUS or other phases of the CTA but negative on CTA in the delayed phase, we will compute Clopper Pearson Exact 95% confidence interval since such a rate could be small. To assess consistency of endoleak type (type 1-5) between CEUS and delayed phase CTA, Kappa coefficient will be used. In the situation with high agreement biased towards one endoleak type, or extremely unbalanced distribution of endoleak types, prevalence-adjusted bias-adjusted kappa coefficient (PABAK) (Byrt, Bishop, and Carlin 1993) will be used. The discrepancy of endoleak type between CEUS and delayed phase CTA will be reported as rate, for example percent of case rated as type 1 in CTA but type 2 in delayed phase, with Clopper Pearson Exact 95% confidence interval. SAS9.4 will be used for all statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 18 or over 2. Able to give informed consent 3. Undergone an EVAR or FEVAR for abdominal aortic aneurysms 4. Expected to have CTA

Exclusion Criteria:

* Unable to receive CTA (Contrast Allergy, Insufficient renal function for standard outpatient contrast study (eGFR <30) Overactive thyroid gland)
* Unable to receive CEUS contrast, previous reaction to Ultrasound Contrast Agent (UCA)
* BMI >50

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
To determine the sensitivity and specificity for CEUS and various CTA phases when using delay phase of CTA as the gold standard | 24 months
  Binomial 95% confidence interval will be calculated for sensitivity and specificity. One- sided binomial test will be conducted to test whether the target sensitivity and specificity are superior to the null value, e.g. a minimal acceptable level of sensitivity and specificity.
Is there any endoleak positive on CEUS or various phases of the CTA but negative on CTA in the delayed phase | 24 months
  In detecting the rate of endoleak positive on CEUS or other phases of the CTA but negative on CTA in the delayed phase, we will compute Clopper Pearson Exact 95% confidence interval since such a rate could be small. To assess consistency of endoleak type (type 1-5) between CEUS and delayed phase CTA, Kappa coefficient will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Grant, Principal Investigator — University of Southern California
Locations (1):
- USC Department of Radiology, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No